CLINICAL TRIAL: NCT02680600
Title: Pharmacokinetic Evaluation of Cefepime Administrered Intravenously in Intensive Care Patients
Brief Title: Individualized Cefepime Dosing Study
Acronym: INCED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Onze Lieve Vrouw Hospital (Other)
Collaborators: University Ghent (Other)
Responsible Party: Principal Investigator, Stijn Jonckheere, Principal Investigator, Onze Lieve Vrouw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B126201419859
Record Dates: First submitted 2016-02-06; First posted 2016-02-11 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Antimicrobial Treatment
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study arm (Experimental): * Cefepime dosing
  * Blood sampling
  * Urine sampling
  * Determination of renal markers
  * Population pharmacokinetic modeling
  * Covariate screening
  * Monte Carlo simulations
  Interventions: Drug: Cefepime dosing; Other: Blood sampling; Other: Urine sampling; Other: Determination of renal markers; Other: Population pharmacokinetic modeling; Other: Covariate screening; Other: Monte Carlo simulations

INTERVENTIONS:
Drug: Cefepime dosing — Patients will received cefepime administered per standard-of-care as a 30 min intravenous infusion. Dosing will be based on local guidelines (the Sanford guide to antimicrobial therapy 2012-2013) using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine formula to estimate glomerular filtration rate (GFR).
  Other Names: Cefepime administration
Other: Blood sampling — Blood will be sampled immediately prior to dose administration (time = 0 at the start of the 30 min infusion), at 0.5, 1, 3, 5 hours post-start of infusion and just before the subsequent dose. From day two onwards, samples will be taken at the end of the infusion and just before the next dose. For the quantification of cefepime, a validated solid phase extraction-liquid chromatography electrospray-tandem mass spectrometry method will be used.
Other: Urine sampling — Timed urine collections were taken during one dosing interval (8 hours in a three times daily regimen) every day.
Other: Determination of renal markers — Creatinine (modified Jaffe method) and urea in serum will be determined using an Architect c16000 analyzer (Abbott, Chicago, IL, USA). Cystatin C will be determined using a particle-enhanced immunonephelometric assay (N Latex Cystatin C, Siemens Healthcare Diagnostics, Marburg, Germany) by use of a BN II nephelometer (Siemens Healthcare Diagnostics). This assay has a calibration traceable to the first certified reference material for cystatin C in human serum (ERM-DA471/IFCC). Kidney injury molecule-1 (KIM-1) in urine and uromodulin in serum will be determined using commercially available ELISA assays: Quantikine ELISA Human TIM-1/KIM-1/HAVCR (R&D Systems, Minneapolis, MN, USA) and Uromodulin ELISA (Euroimmun, Luebeck, Germany), respectively.
Other: Population pharmacokinetic modeling — The cefepime concentration versus time data will be fitted using the FOCE-I estimation algorithm in NONMEM® (Version 7.3; GloboMax LLC, Hanover, MD, USA). R® (R foundation for statistical computing, Vienna, Austria) will be used to graphically assess the model's goodness-of-fit and to evaluate the model's predictive capabilities. As a measure of prediction error, the absolute prediction error (APE) will be used. In short, the measured cefepime concentrations for each individual i at time point j were compared against the population predicted cefepime concentrations, i.e. the predictions for each individual without taking into account the between-subject variability (PRED in NONMEM). The distribution of APEs will be summarized by the median and 90% percentile.
Other: Covariate screening — Renal function will be assessed by four serum based kidney markers (serum creatinine, cystatin C, urea and uromodulin) and two urinary markers (measured creatinine clearance (CrCl) and KIM-1, both on timed urine collections). Serum creatinine and cystatin C will also be used to calculate the eGFR based on CKD-EPI formulas.
Other: Monte Carlo simulations — Based on the final covariate model, a Monte Carlo-based simulation study will be performed to evaluate the Sanford dose recommendations for ICU patients.

SUMMARY:
Several population pharmacokinetic (PK) models for cefepime in critically ill patients have been described, all indicating that variability in renal clearance is the main determinant of observed variability in exposure. The main objective of this study was hence to determine which renal marker best predicts cefepime clearance.

DETAILED DESCRIPTION:
Timely and appropriate antibiotic therapy, sufficient to guarantee adequate antibiotic concentrations in blood and tissues, is one of the most important interventions in critically ill patients with infections.1,2 Cefepime is a fourth generation cephalosporin with broad spectrum activity against Gram-negative bacteria that is used as empirical and directed therapy for severe infections like sepsis and pneumonia. Nevertheless, administration of adequate antibiotic doses is a real challenge in critically ill patients because the pharmacokinetics (PK) of these drugs may be influenced by the complex pathophysiological changes that occur during sepsis.2 Recent reviews described the enormous pharmacokinetic variability of beta-lactam antibiotics in critically ill patients.3,4 Therefore, strategies for dose individualization are explored in an attempt to better control a patient's exposure to the antibiotic, thereby potentially improving the prognosis of critically ill patients with infection. On the one hand, several smaller studies have already shown that better outcomes for critically ill patients can be expected with higher drug exposures, at least for less severely ill patients.5,6 This conclusion was supported by the DALI study, a large multi-center prospective study.7 On the other hand, it was shown that insufficient antibiotic exposure may lead to the development of antibiotic resistance.8 This link was initially shown with inappropriately low quinolone exposures, but more recently with other classes of antibiotics including beta-lactams.9,10 In addition to ensuring that plasma levels are high enough for optimal antimicrobial activity and suppressing emergence of resistance, individualized dosing might offer a perspective to prevent potential side-effects originating from toxic plasma levels. This seems particularly relevant for cefepime, a beta-lactam antibiotic, as it was shown that cefepime is an underappreciated cause of neurotoxicity, especially in intensive care unit (ICU) patients,11,12 patients with impaired renal function,13-16 and patients with brain disorders.17 Population pharmacokinetic models provide a quantitative view of the effect of particular individual factors on the plasma concentration time profile of a drug. Population PK models thereby help to establish individual treatment regimen in patients, depending on the specific patient covariates that were included in the model. As cefepime is a hydrophilic compound, drug elimination is mainly determined by renal clearance and to a lesser extent by non-renal clearance. Therefore, renal markers have been explored as the main determinant to predict cefepime variability in population PK models.18-24 However, none of the published PK models was developed using both plasma and urinary data, though having access to both matrices may be an advantage to identify clinically relevant covariates. Moreover, only creatinine-based markers were used as covariates and, up to now, it was unclear whether the newer markers to assess renal function (e.g. cystatine C, uromodulin and Kidney Injury Moleclure-1 (KIM-1)) are more accurate to predict cefepime clearance.

In this study, a clinical trial was conducted to develop a population PK model for cefepime in critically ill patients assessing renal and non-renal clearance separately, based on both plasma and urinary cefepime concentrations. This model then served as a tool to compare the adequacy of six different renal markers as predictors for renal cefepime clearance. After integrating the most adequate predictor into the PK model, the final model was used to evaluate current dose recommendations for cefepime.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 years or more
* Hospitalized in the ICU of OLV hospital Aalst
* Elected by the treating physician to receive cefepime,irrespectively of the study
* Presence of arterial or central line for blood sampling

Exclusion Criteria:

* Exact time of cefepime administration or blood sampling unknown
* No written informed consent by the patient or his/her (legal) representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Median absolute predictive error (MdAPE) of population PK model without covariates | Evaluation during a maximum follow-up period of 5 days
Median absolute predictive error (MdAPE) of population PK model with different renal markers incorporated | Evaluation during a maximum follow-up period of 5 days

SECONDARY OUTCOMES:
The estimated probability of target attianment (%) for the different categories of the Sanford guide | Based on data from a maximum follow-up period of 5 days
The estimated probability of toxic levels (%) for the different categories of the Sanford guide | Based on data from a maximum follow-up period of 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Stijn Jonckheere, Principal Investigator — Onze Lieve Vrouw Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb SA, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including the Pediatric Subgroup. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Crit Care Med. 2013 Feb;41(2):580-637. doi: 10.1097/CCM.0b013e31827e83af. PMID 23353941
- [Background] Roberts JA, Lipman J. Pharmacokinetic issues for antibiotics in the critically ill patient. Crit Care Med. 2009 Mar;37(3):840-51; quiz 859. doi: 10.1097/CCM.0b013e3181961bff. PMID 19237886
- [Background] Goncalves-Pereira J, Povoa P. Antibiotics in critically ill patients: a systematic review of the pharmacokinetics of beta-lactams. Crit Care. 2011;15(5):R206. doi: 10.1186/cc10441. Epub 2011 Sep 13. PMID 21914174
- [Background] Sime FB, Roberts MS, Peake SL, Lipman J, Roberts JA. Does Beta-lactam Pharmacokinetic Variability in Critically Ill Patients Justify Therapeutic Drug Monitoring? A Systematic Review. Ann Intensive Care. 2012 Jul 28;2(1):35. doi: 10.1186/2110-5820-2-35. PMID 22839761
- [Background] Li C, Du X, Kuti JL, Nicolau DP. Clinical pharmacodynamics of meropenem in patients with lower respiratory tract infections. Antimicrob Agents Chemother. 2007 May;51(5):1725-30. doi: 10.1128/AAC.00294-06. Epub 2007 Feb 16. PMID 17307978
- [Background] McKinnon PS, Paladino JA, Schentag JJ. Evaluation of area under the inhibitory curve (AUIC) and time above the minimum inhibitory concentration (T>MIC) as predictors of outcome for cefepime and ceftazidime in serious bacterial infections. Int J Antimicrob Agents. 2008 Apr;31(4):345-51. doi: 10.1016/j.ijantimicag.2007.12.009. Epub 2008 Mar 4. PMID 18313273
- [Background] Roberts JA, Paul SK, Akova M, Bassetti M, De Waele JJ, Dimopoulos G, Kaukonen KM, Koulenti D, Martin C, Montravers P, Rello J, Rhodes A, Starr T, Wallis SC, Lipman J; DALI Study. DALI: defining antibiotic levels in intensive care unit patients: are current beta-lactam antibiotic doses sufficient for critically ill patients? Clin Infect Dis. 2014 Apr;58(8):1072-83. doi: 10.1093/cid/ciu027. Epub 2014 Jan 14. PMID 24429437
- [Background] Roberts JA, Kruger P, Paterson DL, Lipman J. Antibiotic resistance--what's dosing got to do with it? Crit Care Med. 2008 Aug;36(8):2433-40. doi: 10.1097/CCM.0b013e318180fe62. PMID 18596628
- [Background] Fantin B, Farinotti R, Thabaut A, Carbon C. Conditions for the emergence of resistance to cefpirome and ceftazidime in experimental endocarditis due to Pseudomonas aeruginosa. J Antimicrob Chemother. 1994 Mar;33(3):563-9. doi: 10.1093/jac/33.3.563. PMID 8040120
- [Background] Gugel J, Dos Santos Pereira A, Pignatari AC, Gales AC. beta-Lactam MICs correlate poorly with mutant prevention concentrations for clinical isolates of Acinetobacter spp. and Pseudomonas aeruginosa. Antimicrob Agents Chemother. 2006 Jun;50(6):2276-7. doi: 10.1128/AAC.00144-06. No abstract available. PMID 16723607
- [Background] Fugate JE, Kalimullah EA, Hocker SE, Clark SL, Wijdicks EF, Rabinstein AA. Cefepime neurotoxicity in the intensive care unit: a cause of severe, underappreciated encephalopathy. Crit Care. 2013 Nov 7;17(6):R264. doi: 10.1186/cc13094. PMID 24200036
- [Background] Beumier M, Casu GS, Hites M, Wolff F, Cotton F, Vincent JL, Jacobs F, Taccone FS. Elevated beta-lactam concentrations associated with neurological deterioration in ICU septic patients. Minerva Anestesiol. 2015 May;81(5):497-506. Epub 2014 Sep 15. PMID 25220556
- [Background] Mani LY, Kissling S, Viceic D, Vogt B, Burnier M, Buclin T, Renard D. Intermittent hemodialysis treatment in cefepime-induced neurotoxicity: case report, pharmacokinetic modeling, and review of the literature. Hemodial Int. 2015 Apr;19(2):333-43. doi: 10.1111/hdi.12198. Epub 2014 Jul 23. PMID 25052578
- [Background] Kim A, Kim JE, Paek YM, Hong KS, Cho YJ, Cho JY, Park HK, Koo HK, Song P. Cefepime- Induced Non-Convulsive Status Epilepticus (NCSE). J Epilepsy Res. 2013 Jun 30;3(1):39-41. doi: 10.14581/jer.13008. eCollection 2013 Jun. PMID 24649471
- [Background] Durand-Maugard C, Lemaire-Hurtel AS, Gras-Champel V, Hary L, Maizel J, Prud'homme-Bernardy A, Andrejak C, Andrejak M. Blood and CSF monitoring of cefepime-induced neurotoxicity: nine case reports. J Antimicrob Chemother. 2012 May;67(5):1297-9. doi: 10.1093/jac/dks012. Epub 2012 Jan 31. No abstract available. PMID 22298349
- [Background] Gangireddy VG, Mitchell LC, Coleman T. Cefepime neurotoxicity despite renal adjusted dosing. Scand J Infect Dis. 2011 Oct;43(10):827-9. doi: 10.3109/00365548.2011.581308. Epub 2011 May 23. PMID 21604923
- [Background] Tanaka A, Takechi K, Watanabe S, Tanaka M, Suemaru K, Araki H. Comparison of the prevalence of convulsions associated with the use of cefepime and meropenem. Int J Clin Pharm. 2013 Oct;35(5):683-7. doi: 10.1007/s11096-013-9799-3. Epub 2013 Jun 4. PMID 23733559
- [Background] Lipman J, Wallis SC, Boots RJ. Cefepime versus cefpirome: the importance of creatinine clearance. Anesth Analg. 2003 Oct;97(4):1149-1154. doi: 10.1213/01.ANE.0000077077.54084.B0. PMID 14500173
- [Background] Tam VH, McKinnon PS, Akins RL, Drusano GL, Rybak MJ. Pharmacokinetics and pharmacodynamics of cefepime in patients with various degrees of renal function. Antimicrob Agents Chemother. 2003 Jun;47(6):1853-61. doi: 10.1128/AAC.47.6.1853-1861.2003. PMID 12760858
- [Background] Roos JF, Bulitta J, Lipman J, Kirkpatrick CM. Pharmacokinetic-pharmacodynamic rationale for cefepime dosing regimens in intensive care units. J Antimicrob Chemother. 2006 Nov;58(5):987-93. doi: 10.1093/jac/dkl349. Epub 2006 Aug 30. PMID 16943209
- [Background] Georges B, Conil JM, Seguin T, Dieye E, Cougot P, Decun JF, Lavit M, Samii K, Houin G, Saivin S. Cefepime in intensive care unit patients: validation of a population pharmacokinetic approach and influence of covariables. Int J Clin Pharmacol Ther. 2008 Apr;46(4):157-64. doi: 10.5414/cpp46157. PMID 18397688
- [Background] Delattre IK, Musuamba FT, Jacqmin P, Taccone FS, Laterre PF, Verbeeck RK, Jacobs F, Wallemacq P. Population pharmacokinetics of four beta-lactams in critically ill septic patients comedicated with amikacin. Clin Biochem. 2012 Jul;45(10-11):780-6. doi: 10.1016/j.clinbiochem.2012.03.030. Epub 2012 Apr 5. PMID 22503878
- [Background] Nicasio AM, Ariano RE, Zelenitsky SA, Kim A, Crandon JL, Kuti JL, Nicolau DP. Population pharmacokinetics of high-dose, prolonged-infusion cefepime in adult critically ill patients with ventilator-associated pneumonia. Antimicrob Agents Chemother. 2009 Apr;53(4):1476-81. doi: 10.1128/AAC.01141-08. Epub 2009 Feb 2. PMID 19188394
- [Background] Lima-Rogel V, Medina-Rojas EL, Del Carmen Milan-Segovia R, Noyola DE, Nieto-Aguirre K, Lopez-Delarosa A, Romano-Moreno S. Population pharmacokinetics of cefepime in neonates with severe nosocomial infections. J Clin Pharm Ther. 2008 Jun;33(3):295-306. doi: 10.1111/j.1365-2710.2008.00913.x. PMID 18452417